CLINICAL TRIAL: NCT04348422
Title: Evaluation of the Immune Response in Symptomatic and Asymptomatic Patients' Diagnosed Witih COVID-19
Brief Title: Evaluating the Immune Response for COVID-19
Acronym: COVIDIMMUNE
Status: Completed | Type: Observational
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Principal Investigator, Prof. Shay Efrati, Head of Research and Development Unit, Shamir Medical Center, Assaf-Harofeh Medical Center
Other Study IDs: 105-20-ASF
Record Dates: First submitted 2020-04-13; First posted 2020-04-16 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Nucleic Acid Testing; COVID-19 Serological Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Nasoropharyngeal swabs Blood samples for serology: IgM, IgG, IgA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Symptomatic: COVID-19 RT-PCR positive patients with reported symptoms
  Interventions: Diagnostic Test: COVID-19 RT-PCR; Diagnostic Test: COVID-19 Serology; Other: Symptoms questionnare
- Asymptomatic: COVID-19 RT-PCR positive patients without presenting any symptoms
  Interventions: Diagnostic Test: COVID-19 RT-PCR; Diagnostic Test: COVID-19 Serology; Other: Symptoms questionnare

INTERVENTIONS:
Diagnostic Test: COVID-19 RT-PCR — Nasoropharyngeal swabs for COVID-19 RT-PCR - initial screening/retest +every 10 days in 100 days followup period
Diagnostic Test: COVID-19 Serology — Blood samples for COVID-19 serology - initial screening/retest +every 10 days in 100 days followup period Each sample will be examined by 4-6 serology kits.
Other: Symptoms questionnare — Symptoms questionnaire which will be filled by participant on initial screening/retest visit + every 10 days in 100 days followup period

SUMMARY:
The 2019-20 coronavirus disease, caused by COVID-19, is an ongoing pandemic. The measures in which public health officials quarantine confirmed and isolate symptomatic cases in order to reduce the spread COVID-19 is the common practice used in most countries. However, a significant question remains in regards to the asymptomatically infected individuals, which may propagate the virus and impede infection control. The other question to consider is whether these asymptomatic carriers develop an immune response or continue viral shedding. The purpose of the current study is the evaluate the immune response, i.e developing anti-SARS-CoV-2 antibodies in the asymptomatic cases, in a household study design.

We plan to evaluate over 1000 patients with positive COVID-19 results and their households.

DETAILED DESCRIPTION:
The 2019-20 coronavirus disease, caused by COVID-19, is an ongoing pandemic. The outbreak started in Wuhan, Hubei province, China, in December 2019 and the World Health Organization (WHO) recognized it as a pandemic on 11 March 2020. Up to Apr 9. 2020 there are more than 1.4 million confirmed cases, and over 82,000 deaths 1. In Israel, COVID-19 was confirmed in more 9,000 cases and took the life of 70 victims (09.04.2020) .

With the extensive outbreak of COVID-19, a mass of studies with a large population have been reported. Wu et al. found that the mean R0 of COVID-19 was approximately 2.68(95% CI: 2.47-2.86) . The measures in which public health officials quarantine confirmed and isolate symptomatic cases in order to reduce the spread COVID-19 is the common practice used in most countries. However, a significant question remains in regards to the asymptomatically infected individuals, which may propagate the virus and impede infection control.

The problem To date, initial surveillance has focused primarily on patients with severe disease, and, as such, the full spectrum of the disease. The extent of asymptomatic disease is not clear. Mizumoto et al. mathematical model suggested 17.9-33.3% are asymptomatic carriers. The other question to consider is whether these asymptomatic carriers develop an immune response or continue viral shedding.

SARS-CoV-2, the causative viral agent of the disease COVID-19, is a coronavirus which bears the transmembrane glycoprotein spikes (S protein) typical of viruses in its clade. The spikes on SARS-CoV-2 allows the virus to enter host cells through the human receptor angiotensin converting enzyme 2 (ACE2), present in alveolar epithelial cells. These spikes are a prominent target of human immune responses and have been found to be highly immunogenic and induce antibody production. The receptor-binding domain (RBD) of the S protein is particularly targeted by neutralizing antibodies.

The diagnostic test in symptomatic patients is based on real time polymerase chain reaction (RT-PCR), which tests the existence of specific COVID-19 genes in the sample. However, there are growing numbers of reports of false negative results due to improper sample collection, low viral load or technical instability of the PCR.

Serology test aims to detect antibodies (immunoglobulin M - IgM, immunoglobulin G- IgG, immunoglobulin A - IgA) in the patient's' blood, i.e. the patient's immune response. The IgM antibodies usually show within 3-7 days from symptoms, whereas IgG antibodies follow within 10-14 days. Diseases which involve the respiratory tract usually cause elevation of IgA as well.

Zhao et al. have recently published data indicating that COVID-19 patients show typical antibody production times in response to acute viral infection with SARS-CoV-2. Overall, the data suggest that SARS-CoV-2 infection follows a seroconversion timeline similar to other viral infections. In their sample of 173 of hospitalized symptomatic confirmed patients, 93.1% (161/173) developed antibodies, where 82.7% developed IgM antibodies and 64.7% developed IgG antibodies. Importantly, all of these patients suffered from symptoms. The association between symptoms level, viral load and the immune response is yet to be determined.

Closed settings, such as households, have a defined population that may not mix readily with the larger surrounding community, and therefore such settings can provide a strategic way to track emerging respiratory infections and characterize virus transmission patterns because the denominator can be well defined. Also, exposure is within the setting, and follow-up of household contacts is generally more feasible in this well-defined setting as compared to an undefined one. Following close contacts with similar levels of exposure to infection from primary cases can also permit identification of the asymptomatic fraction.

Our solution The purpose of the current study is the evaluate the immune response, i.e developing anti-SARS-CoV-2 antibodies in the asymptomatic cases, in a household study design.

We plan to evaluate over 1000 patients with positive COVID-19 results and their households. The plan includes evaluation of their symptoms, viral load and immune response every 10 days in a period of 12 weeks. Next, Analysis of the cause of the immune response differences between subjects by sequencing their DNA and most importantly of the ACE2 gene - the receptor the virus attacks.

This will shed the needed light on the connection between symptoms, viral load and immune response. The association between viral load, symptoms and immune response will enable: monitor disease progress, predict patients who are at high risk to develop severe symptoms, determine immunity to the virus and most importantly locate the chronic carriers which do not develop immunity.

Protocol Following a positive COVID-19 RT-PCR result in the Shamir medical center lab, the subject will be contacted by telephone and will be offered to participate in the study. Upon consent, medical staff will arrive to the subject's house and further explain the details of the study and ask for an informed consent of the subject and any of the households over 18 years old. Upon signing an informed consent, each of the subject will fill a symptoms report and provide an oropharyngeal swab and blood sample (10-20cc).

Every 10 days within 12 weeks, a researcher will visit the subjects house, and repeat the procedure (symptoms questionnaire, blood withdrawal and oropharyngeal swab).

Following the last evaluation (12th week), every 4-8 weeks within 1 year, a researcher will visit the subjects hosue and perform filling of symptoms questionnaire and blood withdrawal.

Serology kits:

1. LIAISION SARS-CoV-2 IgM (Diasorin, Saluggia, Italy)
2. LIAISION SARS-CoV-2 S1/S2 IgG (Diasorin, Saluggia, Italy)
3. ARCHITECT SARS-CoV-2 N IgG Immunoassay (Abbot, Illinois, U.S.A)

Rt-PCR kit RT-PCR will be performed using 3 primers and 3 probes in addition to one human RNase primer and probe.

Procedure

1. Arrival to the subjects house
2. Medical staff will use appropriate protective medical gear.
3. Blood withdrawal for 3 blood tubes (15-20cc)
4. Oropharyngeal swab
5. Samples will be kept at 2-8c degrees.
6. Samples will be returned to Shamir Medical Center lab in 2-8c degrees.
7. RT-PCR will be performed.
8. Serology will be performed using the available kits. Each subject will be sampled 9 times (every 10 days within 12 weeks in addition to the first contact). Blood samples will be kept and stored at -80°C for future research purposes.

Long term evaluation will include Blood sample and questionnaires every 4-8 weeks for 1 year from the final evaluation (12th week).

Timing

1. The first evaluation will be completed for both the patient and his/her households within 1-7 days of receiving the RT-PCR positive result
2. Following the first evaluation, each participant will be evaluated every 10 days (±2 days) for 100 days. In total 10 additional times.

   In summary, each participant will be evaluated 11 times (first evaluation + 10 additional evaluations).
3. Following the last evaluation, each participant will be evaluated every 4-8 weeks for 1 year. In total 6-12 times.

ELIGIBILITY:
Inclusion Criteria:

* Positive COVID-19 RT-PCR to the subject or his/her household.
* Over 18 years old
* Ability to sign an informed consent

Exclusion Criteria:

* Inability to sign an informed consent
* Pregnancy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who were found positive in a clinical RT-PCR diagnostic test in the Shamir Medical Center and their households.
  Following a positive COVID-19 RT-PCR result in the Shamir medical center lab, the subject will be contacted by telephone and will be offered to participate in the study. Upon consent, medical staff will arrive to the subject's house and further explain the details of the study and ask for an informed consent of the subject and any of the households over 18 years old.
Sampling Method: Non-Probability Sample
Enrollment: 214 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2022-02-02 (Actual); Study Completion 2022-02-02 (Actual)

PRIMARY OUTCOMES:
Proportion of symptomatic patients with immune response (IgM/IgG/IgA) | 100 days
  The percentage of symptomatic patients who developed either IgM/IgG/IgA response within 100 days from COVID-19 Infection
Proportion of Asymptomatic patients with immune response (IgM/IgG/IgA) | 100 days
  The percentage of Asymptomatic patients who developed either IgM/IgG/IgA response within 100 days from COVID-19 Infection

SECONDARY OUTCOMES:
Time to IgM | Evaluated within a 100 days followup
  the mean time patients devleoped IgM
Time to IgG | Evaluated within a 100 days followup
  the mean time patients devleoped IgG
Time to IgA | Evaluated within a 100 days followup
  the mean time patients devleoped IgG
Serology kits inter-observer agreement | Evaluated within a 100 days followup
  Cohen's kappa coefficient calculated between the different serology kits used for evaluation
Proportion of symptomatic patients with immune response (IgM/IgG/IgA)- long term | 1 year
  The percentage of symptomatic patients who developed either IgM/IgG/IgA response within 1-1.3 years from COVID-19 Infection
Proportion of Asymptomatic patients with immune response (IgM/IgG/IgA) -long term | 1 year
  The percentage of symptomatic patients who developed either IgM/IgG/IgA response within 1-1.3 years from COVID-19 Infection

CONTACTS AND LOCATIONS:
Overall Officials: Shai Efrati, MD, Principal Investigator — Head of Research and Development Unit
Locations (1):
- Assaf-Harofeh Medical Center, Ramla, Israel

IPD SHARING:
Plan to Share IPD: Undecided
Anonymous data may be shared upon request

REFERENCES:
- [Background] Wu JT, Leung K, Leung GM. Nowcasting and forecasting the potential domestic and international spread of the 2019-nCoV outbreak originating in Wuhan, China: a modelling study. Lancet. 2020 Feb 29;395(10225):689-697. doi: 10.1016/S0140-6736(20)30260-9. Epub 2020 Jan 31. PMID 32014114
- [Background] Bai Y, Yao L, Wei T, Tian F, Jin DY, Chen L, Wang M. Presumed Asymptomatic Carrier Transmission of COVID-19. JAMA. 2020 Apr 14;323(14):1406-1407. doi: 10.1001/jama.2020.2565. PMID 32083643
- [Background] Mizumoto K, Kagaya K, Zarebski A, Chowell G. Estimating the asymptomatic proportion of coronavirus disease 2019 (COVID-19) cases on board the Diamond Princess cruise ship, Yokohama, Japan, 2020. Euro Surveill. 2020 Mar;25(10):2000180. doi: 10.2807/1560-7917.ES.2020.25.10.2000180. PMID 32183930
- [Background] Zhao J, Yuan Q, Wang H, Liu W, Liao X, Su Y, Wang X, Yuan J, Li T, Li J, Qian S, Hong C, Wang F, Liu Y, Wang Z, He Q, Li Z, He B, Zhang T, Fu Y, Ge S, Liu L, Zhang J, Xia N, Zhang Z. Antibody Responses to SARS-CoV-2 in Patients With Novel Coronavirus Disease 2019. Clin Infect Dis. 2020 Nov 19;71(16):2027-2034. doi: 10.1093/cid/ciaa344. PMID 32221519
- See also: WHO COVID-19 situation reports — https://www.who.int/emergencies/diseases/novel-coronavirus-2019/situation-reports